CLINICAL TRIAL: NCT05321043
Title: Risk Assessment of Indirect Exposure to the Environment in the Gastrointestinal Endoscopy Center
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Tsinghua University (Other)
Responsible Party: Principal Investigator, SHENGYU ZHANG, Associate Professor, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ZS-3367
Record Dates: First submitted 2022-03-16; First posted 2022-04-11 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Infection Control
Keywords: infection control; indirect contagion transmission; digestive endoscopy center

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vitamin B2 labeled group (Other): A liquid of vitamin B2 and hand sanitizer (0.12mg/mL) is marked on the patients' hands outside the endoscopy center.
  Interventions: Other: Vitamin B2 labeling

INTERVENTIONS:
Other: Vitamin B2 labeling — Using medical non-toxic fluorescent agents, VB2 solution, to mark the patient's hands before endoscopy examination.

SUMMARY:
Study objective: To clarify the risk of exposure to indirect contact and transmission of environmental objects during digestive endoscopy diagnosis and treatment for patients and medical staff, simulating by using Vitamin B2 solution.

Study design: This is a case-only research.

DETAILED DESCRIPTION:
In the study, the object surface of the digestive endoscopy room is preliminarily analyzed, and several key exposure units, such as potential high-frequency touch areas such as the surface of the bed unit, are screened and defined. A fluorescence photographing system is arranged in the digestive endoscopy room, and the exposure unit before treatment is photographed with the best excitation wavelength of the fluorescent marker as the light source, to get the experimental background reference. Then, patients undergoing digestive endoscopy in the same endoscopy work unit (usually half a day) are selected. Before entering the digestive center, the hands of patients are fluorescently marked with vitamin B2 mixed hand sanitizer 1ml (vitamin B2 0.12mg/ml). Meanwhile, the process of the gastroscopy is recorded by camera for the recognition of touch behaviors. Then, the doctors and nurses give routine care and procedure. Based on the fluorescence tracing and detection methods, the indoor light source is turned off after each selected endoscopy work unit, and the fluorescence residue on the surface of key exposed units is photographed. The environmental surfaces touched by the patient are sampled by the wiping method. Then the video of the gastroscopy process is analyzed for the recognition of touch behaviors. The dosage is detected by the Fluoro Max-4® fluorophotometer (HORIBA, Japan), which is quantified as a cumulative mass (μg) over all the exposure time.

ELIGIBILITY:
Inclusion Criteria:

* During the study period, patients who were treated in the digestive endoscopy center of Beijing Union Medical College Hospital and planned to undergo gastroscopy. Age and gender are not limited temporarily.

Exclusion Criteria:

* Allergic to medical non-toxic fluorescent agent: Vitamin B2 aqueous solution.
* Poor general condition, including severe cardiopulmonary disease, difficult to tolerate examination, and coagulation disorders.
* Patients with contraindications to endoscopy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Dosage of Indirect Contact Exposure of Environmental surfaces | one year
  A liquid of Vitamin B2 and hand sanitizer (0.12mg/mL) is marked on the hands of every patient who is scheduled in the same endoscopy work unit (usually half a day) outside the endoscopy center. Then, the doctors and nurses conduct standard EGD procedure. After this endoscopy work unit is finished, the environmental surfaces touched by the patient are sampled by the wiping method. The dosage is detected by the Fluoro Max-4® fluorophotometer (HORIBA, Japan), which is quantified as a cumulative mass (μg) over all the exposure time.

CONTACTS AND LOCATIONS:
Overall Officials: Shengyu Zhang, MD, Study Director — Peking Union Medical College Hospital; Yuheng Zhang, MD candidate, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China